CLINICAL TRIAL: NCT00465218
Title: "Transcranial Doppler Assessment of Cerebral Embolization During Early Anti-thrombotic Therapy After Bioprosthetic Aortic Valve Replacement: Comparison of High-dose Aspirin Versus Warfarin Plus Low-dose Aspirin"
Brief Title: Transcranial Doppler (TCD) Assessment During Early Anti-thrombotic Therapy After Bioprosthetic Aortic Valve Replacement
Acronym: Tissue-Valve
Status: Completed | Type: Observational
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Principal Investigator, Marc Ruel MD MPH FRCSC, Dr., Ottawa Heart Institute Research Corporation
Other Study IDs: 2006785-01H
Record Dates: First submitted 2007-04-20; First posted 2007-04-24 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Aortic Valve Disease
Keywords: Bioprosthesis; Thrombosis; Cerebral emboli; Transcranial Doppler; Platelet function tests
MeSH Terms: conditions — Aortic Valve Disease; Thrombosis; Intracranial Embolism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: High dose aspirin (325 mg)
  Interventions: Procedure: Prophylaxis of Thrombosis after aortic valve replacement
- 2: Low dose aspirin (81 mgs) plus warfarin
  Interventions: Procedure: Prophylaxis of Thrombosis after aortic valve replacement

INTERVENTIONS:
Procedure: Prophylaxis of Thrombosis after aortic valve replacement — Two standard prophylactic treatments of thrombosis within the first 3 months postsurgery currently used in our institution: a) daily dose of aspirin (325 mgs; b) daily dose of aspirin (81 mg) plus Warfarin for target INR 2.0-2.5

SUMMARY:
The purpose of this study is to determine if there is any difference in the counts of cerebral emboli and platelet function between two prophylactic treatments of thrombosis currently used at University of Ottawa Heart Institute for the first three months after surgery in low-risk patients undergoing aortic valve replacement with a bioprosthetic valve: 1) daily use of high-dose aspirin [325 mgs], and 2) the combination of oral Warfarin [target INR 2.0 to 3.0] and low-dose aspirin [81 mg].

DETAILED DESCRIPTION:
Background:

There are several medications used to prevent blood clotting in patients undergoing surgical replacement of their aortic valves with tissue valves. One of these medications is called warfarin (Coumadin ®) which prevents blood clotting by making the blood "thinner." Another medication is aspirin which prevents the aggregation (clustering) of cells in the blood called platelets. Some clinicians consider that using only aspirin should be enough to protect the patients against the presence of clots in the blood, but others consider that aspirin should be combined with warfarin for better protection. Moreover, physicians express concern over the use of oral anticoagulation due to the possibility of an increased risk of bleeding. The effects of these medications for preventing blood clots traveling to the brain after the surgery are currently unknown. Transcranial doppler ultrasound will be used in these patients to evaluate non-invasively the quantity of fragments of clots circulating in the arteries of the brain. In addition, platelet function will be measured to determine how effective these treatments are for preventing the aggregation of the blood cells called platelets, which may be involved in clot formation.

Objective:

Our purpose is to determine if there is any difference in the counts of cerebral emboli and platelet function between two prophylactic treatments of thrombosis currently used in our institution for the first three months after surgery in these patients: 1) daily use of high-dose aspirin [325 mgs], and 2) the combination of oral Warfarin [target INR 2.0 to 3.0] and low-dose aspirin [81 mg].

Methods:

Patients with low risk profile undergoing primary aortic valve replacement with a bioprosthetic (tissue) valve will be eligible for the study. Patients will receive one of the two prophylactic treatments of thrombosis (1 or 2) depending on the surgeon's preference. Platelet function will be measured before surgery and transcranial doppler within the first 24 hours immediately after the surgery. At the end of one month following surgery, all patients will undergo transcranial doppler and platelet function assessment. The study will be powered on demonstrating the hypothesis of substantial equivalence between the two treatments as regarding the primary outcome (cerebral emboli).

Outcome measures:

1. Primary outcome:

   Bilateral counts of cerebral emboli in the middle cerebral arteries with transcranial doppler ultrasound at one month after surgery
2. Secondary outcomes:

Platelet function, incidence of major adverse neurologic and bleeding events at one month following surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary aortic valve replacement with bioprosthetic (tissue) valve.

Exclusion Criteria:

* Emergency surgery or redo operations.
* Patients with history of transient ischemic attacks, stroke, or history of carotid stenosis greater than 50% as detected by carotid duplex doppler or angiography.
* Patients with COPD who are CO2 retainers.
* Patients with LV function less than 50%, or enlarged left ventricle greater than 50 mm as detected by echocardiography or previous history of thromboembolism.
* Patients with history of atrial fibrillation or heart rhythm disturbances.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with aortic valve stenosis and/or insuficiency undergoing aortic valve replacement with a bioprosthetic valve (tissue valve).
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2007-03; Primary Completion 2007-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Differences in the rate of doppler-detected cerebral micro emboli between the two prophylactic treatments of thrombosis | 1 month after surgery

SECONDARY OUTCOMES:
Differences in the degree of inhibition of platelet aggregation between the two prophylactic treatments of thrombosis | 1 month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ruel, MD, MPH, Principal Investigator — Ottawa Heart Institute Research Corporation; Thierry Mesana, MD, PhD, Study Director — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Gohlke-Barwolf C, Acar J, Oakley C, Butchart E, Burckhart D, Bodnar E, Hall R, Delahaye JP, Horstkotte D, Kremer R, et al. Guidelines for prevention of thromboembolic events in valvular heart disease. Study Group of the Working Group on Valvular Heart Disease of the European Society of Cardiology. Eur Heart J. 1995 Oct;16(10):1320-30. doi: 10.1093/oxfordjournals.eurheartj.a060739. No abstract available. PMID 8746900
- [Background] ACC/AHA guidelines for the management of patients with valvular heart disease. A report of the American College of Cardiology/American Heart Association. Task Force on Practice Guidelines (Committee on Management of Patients with Valvular Heart Disease). J Am Coll Cardiol. 1998 Nov;32(5):1486-588. doi: 10.1016/s0735-1097(98)00454-9. No abstract available. PMID 9809971
- [Background] Stein PD, Alpert JS, Bussey HI, Dalen JE, Turpie AG. Antithrombotic therapy in patients with mechanical and biological prosthetic heart valves. Chest. 2001 Jan;119(1 Suppl):220S-227S. doi: 10.1378/chest.119.1_suppl.220s. PMID 11157651
- [Background] Kirtane AJ, Rahman AM, Martinezclark P, Jeremias A, Seto TB, Manning WJ. Adherence to American College of Cardiology/American Heart Association guidelines for the management of anticoagulation in patients with mechanical valves undergoing elective outpatient procedures. Am J Cardiol. 2006 Mar 15;97(6):891-3. doi: 10.1016/j.amjcard.2005.09.139. Epub 2006 Feb 2. PMID 16516596
- [Background] Heras M, Chesebro JH, Fuster V, Penny WJ, Grill DE, Bailey KR, Danielson GK, Orszulak TA, Pluth JR, Puga FJ, et al. High risk of thromboemboli early after bioprosthetic cardiac valve replacement. J Am Coll Cardiol. 1995 Apr;25(5):1111-9. doi: 10.1016/0735-1097(94)00563-6. PMID 7897124
- [Background] Moinuddeen K, Quin J, Shaw R, Dewar M, Tellides G, Kopf G, Elefteriades J. Anticoagulation is unnecessary after biological aortic valve replacement. Circulation. 1998 Nov 10;98(19 Suppl):II95-8; discussion II98-9. PMID 9852888
- [Background] Gherli T, Colli A, Fragnito C, Nicolini F, Borrello B, Saccani S, D'Amico R, Beghi C. Comparing warfarin with aspirin after biological aortic valve replacement: a prospective study. Circulation. 2004 Aug 3;110(5):496-500. doi: 10.1161/01.cir.0000137122.95108.52. PMID 15289387
- [Background] Rodriguez RA, Rubens F, Rodriguez CD, Nathan HJ. Sources of variability in the detection of cerebral emboli with transcranial Doppler during cardiac surgery. J Neuroimaging. 2006 Apr;16(2):126-32. doi: 10.1111/j.1552-6569.2006.00035.x. PMID 16629734
- [Background] Zimmermann N, Roussiekan T, Winter J, Kurt M, Gams E, Wenzel F, Hohlfeld T. Platelet inhibition by aspirin after aortic valve replacement. J Thorac Cardiovasc Surg. 2006 Jun;131(6):1392-3. doi: 10.1016/j.jtcvs.2006.01.029. No abstract available. PMID 16733175
- [Background] Geiser T, Sturzenegger M, Genewein U, Haeberli A, Beer JH. Mechanisms of cerebrovascular events as assessed by procoagulant activity, cerebral microemboli, and platelet microparticles in patients with prosthetic heart valves. Stroke. 1998 Sep;29(9):1770-7. doi: 10.1161/01.str.29.9.1770. PMID 9731593
- [Background] Sturzenegger M, Beer JH, Rihs F. Monitoring combined antithrombotic treatments in patients with prosthetic heart valves using transcranial Doppler and coagulation markers. Stroke. 1995 Jan;26(1):63-9. doi: 10.1161/01.str.26.1.63. PMID 7839399
- [Background] Markus HS, Thomson ND, Brown MM. Asymptomatic cerebral embolic signals in symptomatic and asymptomatic carotid artery disease. Brain. 1995 Aug;118 ( Pt 4):1005-11. doi: 10.1093/brain/118.4.1005. PMID 7655877